CLINICAL TRIAL: NCT01752712
Title: Combined Oxytocin and CBSST for Social Function in People With Schizophrenia
Brief Title: Oxytocin and CBSST for People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert Buchanan, Chief, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00054628
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2017-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Oxytocin; Social function; CBSST
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Social Adjustment | interventions — Oxytocin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBSST + oxytocin (Experimental): Cognitive Behavioral Social Skills Training with adjunct oxytocin nasal spray treatment. Participants will receive 80 IU/day of oxytocin administered intranasally in two doses (40 IU morning and evening).
  Interventions: Drug: CBSST + Oxytocin
- CBSST + placebo (Placebo Comparator): Cognitive Behavioral Social Skills Training with placebo nasal spray. The placebo nasal spray bottles will be matched in appearance to the oxytocin nasal spray bottles and similarly administered intranasally in two doses (morning and evening).
  Interventions: Drug: CBSST + Placebo

INTERVENTIONS:
Drug: CBSST + Oxytocin — The oxytocin dose of 80 IU/day, will be administered in two divided doses: 40 IU in the morning and 40 IU in the evening. Oxytocin will be administered intranasally (10 puffs of the spray, 5 in each nostril at each administration). CBSST groups will occur for an hour twice/week. Nasal spray will be administered an hour prior to the CBSST group.
  Arms: CBSST + oxytocin
Drug: CBSST + Placebo — Matching placebo spray will be administered intranasally (10 puffs of the spray, 5 in each nostril at each administration). CBSST groups will occur for an hour twice/week. Nasal spray will be administered an hour prior to the CBSST group.
  Other Names: sugar pill
  Arms: CBSST + placebo

SUMMARY:
A significant proportion of people with schizophrenia are characterized by impaired ability to socially engage with others, which may reflect social aversion secondary to defeatist beliefs; decreased motivation for social interactions; and/or impairment in the normal reinforcement value of social interactions. These impairments in social function have been shown to be associated with social skill deficits; and decreased ability to identify and remember emotional facial expressions and empathize with the emotional status of others. Unfortunately, pharmacological interventions have limited benefits for impaired social function, whereas psychosocial interventions provide only partial benefit for this critical aspect of the illness. The development of an effective intervention for functional outcomes remains a central therapeutic challenge. Cognitive Behavioral Social Skills Training (CBSST) uses corrective feedback and reinforcement provided by successful interactions to challenge and reduce defeatist performance beliefs that contribute to low drive and interfere with social functioning. CBSST has been shown to have modest effects on social function in people with schizophrenia. Oxytocin plays a critical role in the regulation of normal social affiliative behavior; it is hypothesized to enhance social affiliation through the reduction of anxiety or social risk aversion; the enhancement of motivation for prosocial approach behavior; and/or increased modulation of the salience and processing of social cues. People with schizophrenia have decreased oxytocin levels, which are associated with an impaired ability to identify facial emotions and decreased prosocial behaviors. The study will be comprised of three phases: 1) 2-week Evaluation Phase; 2) 24-week Double-blind Treatment Phase; and 3) 3-month Follow-up Phase.

DETAILED DESCRIPTION:
A NIMH mission priority is the development of new and better interventions, whose focus extends beyond symptom amelioration to the development of interventions that allow people who suffer from severe mental illnesses "to live full and productive lives" (NIMH Strategic Plan, 2008). In particular, the NIMH Strategic Plan notes the importance of translating "research on the biological causes of disorder to inform and develop psychosocial and biomedical interventions that target core features of disease, assess outcomes appropriate to the course of illness under study, and develop study designs that have impact on these features." The current proposal is built upon the observations that: 1) people with schizophrenia are characterized by marked impairments in their social function; 2) current pharmacological treatments do not address these impairments; 3) CBSST has been shown to have modest effects on social function in people with schizophrenia. This limited efficacy may be related to the lack of interest or drive people with schizophrenia have for social interactions; 4) oxytocin plays a critical role in normal social affiliative behavior through a) the reduction of anxiety or social risk aversion, b) the enhancement of motivation for prosocial approach or affiliative behavior, and/or c) increased modulation of the salience and processing of social cues; and 5) decreased oxytocin is associated with social function impairments in people with schizophrenia.

The proposed study is based on the proposition that the use of a pharmacological agent, whose behavioral effects compliment the psychological mechanisms of action of a psychosocial intervention, is an important adaptation of an intervention previously shown to have moderate effects on social function. The addition of oxytocin to CBSST is hypothesized to: 1) enhance the reduction of defeatist performance beliefs by reducing social risk aversiveness and avoidance, which would increase exposure to reinforcement and corrective feedback; 2) enhance social skill acquisition through improvement of proximal social behaviors, e.g. making eye contact and attending to the facial expressions of social partners; and 3) facilitate the translation of learned social skills into community practice through its effects on prosocial attachment behaviors, reduction in social disinterest, and effects on distal behaviors, e.g. initiating conversations and responding to social invitations. Increased social risk taking within and between sessions would expose participants to a greater frequency of positive feedback and success experiences, which would provide evidence to dispute their defeatist beliefs and social disinterest attitudes. In addition, increased social risk taking could improve homework adherence (e.g., practicing talking to people in the community) and engagement in new community activities. These interactive effects would subsequently lead to a substantial improvement in CBSST efficacy for social function. Ultimately, the importance of improved social function is the effect that such improvement would have on overall levels of health and functioning, including vocational outcome.

The proposed study will enable us to collect preliminary data on the acceptability, efficacy, feasibility, and safety of the proposed intervention. In particular, this would be the first study to examine the safety of long-term oxytocin in this population. The study will also provide critical data on the feasibility of recruiting and retaining participants with schizophrenia in a long-term intervention, which combines two different therapeutic modalities: CBSST and oxytocin. If found to be efficacious, feasible, and well-tolerated, we will plan to conduct a larger study, which would include the use of cognitive and imaging biomarkers, to more fully elucidate the mechanism of action of the observed treatment effects. The investigators will address the following specific aims:

Aim #1 (Efficacy): To determine if CBSST + oxytocin compared to CBSST + placebo-oxytocin is associated with improved social function.

Aim #2 (Safety): To determine if CBSST + oxytocin compared to CBSST + placebo-oxytocin is associated with increased incidence of side effects.

Aim #3 (Change Mechanism): To determine if CBSST + oxytocin compared to CBSST + placebo-oxytocin is associated with reduced social aversion, including social disinterest and defeatist performance beliefs; increased ability to trust others; and/or improved performance on facial recognition and memory measures.

Aim #4 (Other Outcomes): To determine if CBSST + oxytocin compared to CBSST + placebo-oxytocin is associated with improved neuropsychological test performance, and/or decreased positive, negative, and/or anxiety/depression symptoms, and clinical global improvement.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV-TR diagnosis of schizophrenia or schizoaffective disorder
2. Scale for the Assessment of Negative Symptoms asociality item score ≥ 2
3. Considered clinically stable by the treating psychiatrist
4. Stable treatment with the same antipsychotic for at least 60 days and the same dose for at least the 30 days prior to study entry.
5. Male or female of any race.

Exclusion Criteria:

1. Organic brain disorder, including cerebrovascular accident; epilepsy; traumatic brain injury, loss of consciousness (LOC) for more than 30 minutes
2. Mental retardation
3. Medical conditions, whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol
4. Participant is pregnant or is lactating
5. History of chronic allergic rhinitis
6. DSM-IV-TR diagnosis of alcohol or substance dependence (except nicotine) within the last 6 months, or participant has met dependence criteria for 5 years or more.
7. DSM-IV-TR diagnosis of alcohol or substance abuse (except nicotine) within the last month
8. Participant has a past history of polydypsic hyponatremia (defined by sodium levels below 130 mmol/L) or has a current sodium level below 135 mmol/L
9. Participant with EKG evidence of any of the following cardiac arrhythmias: QTc prolongation (Males: 450 msec or greater; females: 470 msec or greater); atrial fibrillation; ventricular or supraventricular tachycardia; and 2nd or 3rd degree A-V Block

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Buchanan, MD, Principal Investigator — University of Maryland, College Park
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - Maryland Psychiatric Research Center, Baltimore, Maryland

REFERENCES:
- [Derived] Buchanan RW, Kelly DL, Strauss GP, Gold JM, Weiner E, Zaranski J, Chen S, Blatt F, Holden J, Granholm E. Combined Oxytocin and Cognitive Behavioral Social Skills Training for Social Function in People With Schizophrenia. J Clin Psychopharmacol. 2021 May-Jun 01;41(3):236-243. doi: 10.1097/JCP.0000000000001397. PMID 33783399

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 83 participants signed a consent form for the study. 4 of these subjects were deemed ineligible before starting any study procedures, and 17 participants were withdrawn from the study prior to randomization for various reasons. Therefore, 62 subjects were randomized to a study treatment group (31 CBSST+oxytocin, 31 CBSST+placebo).
Period: Overall Study
Arm/Group | CBSST + Oxytocin | CBSST + Placebo
Started | 31 | 31
Completed | 22 | 21
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBSST + Oxytocin | CBSST + Placebo | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (8.7) | 40.7 (10.2) | 41.92 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 18 | 20 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 7 | 16
  White | 17 | 15 | 32
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Birchwood Social Function Scale (BSFS) Total Score
Description: Determine if CBSST + oxytocin compared to CBSST + placebo is associated with improved social function. There are 7 individual sections, with each section asking about different aspects of social functioning. Scores for Section 1: "Social Engagement Withdrawal" range from 0-15; Section 2: "Interpersonal Communication/Relationships" ranges from 0-30; Section 3: "Prosocial Activities" range is 0-66; Section 4: "Recreation" ranges from 0-48; Section 5: "Independence (Performance)" ranges from 0-39; Section 6: "Independence (Competence)" ranges from 0-39; and Section 7: "Occupation/Employment" ranges from 0-6 if the participant is unemployed or 7-10 if the participant is employed. The minimum value possible is 0 for participants who are unemployed and 7 for those with employment. The total BSFS score is calculated by adding the total scores from each of the 7 sections, with a maximum total score of 247. A lower total score indicates a lower social function rating.
Time Frame: Treatment weeks 0, 12, and 24, plus follow-up week 36
Population: Only participants who were enrolled in the study and had completed a BSFS assessment were analyzed at each study time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBSST + Oxytocin | CBSST + Placebo
Number analyzed (Participants) | 31 | 31
units on a scale
  Treatment Week 0 | 120 (23.1) | 115.8 (21.4)
  Treatment Week 12: number analyzed (Participants) | 27 | 25
  Treatment Week 12 | 120.8 (21.9) | 127 (21.8)
  Treatment Week 24: number analyzed (Participants) | 22 | 20
  Treatment Week 24 | 125.3 (20.3) | 126.4 (17.4)
  Follow-Up Week 36: number analyzed (Participants) | 22 | 20
  Follow-Up Week 36 | 124 (20.2) | 125.8 (21.4)

2. Secondary Outcome: Defeatist Performance Attitudes Scale (DPAS) Total Score
Description: Determine if CBSST + oxytocin compared to CBSST + placebo is associated with defeatist performance beliefs. The total DPAS score is calculated by adding the scores for scales #1-#18. Each scale ranges from "1=Agree Totally" to "7=Disagree Totally". Total scores range from a minimum score of 18 to a maximum score of 126. Reverse scoring was applied to make higher scores indicate a stronger defeatist attitude.
Time Frame: Treatment weeks 0, 12, and 24, plus follow-up week 36
Population: Only participants who were enrolled in the study and had completed a DPAS assessment were analyzed at each study time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBSST + Oxytocin | CBSST + Placebo
Number analyzed (Participants) | 31 | 31
units on a scale
  Treatment Week 0 | 68.55 (19.23) | 67.87 (15.31)
  Treatment Week 12: number analyzed (Participants) | 27 | 24
  Treatment Week 12 | 71.22 (19.38) | 66.92 (14.23)
  Treatment Week 24: number analyzed (Participants) | 22 | 20
  Treatment Week 24 | 73.50 (18.07) | 72.65 (16.80)
  Follow-Up Week 36: number analyzed (Participants) | 22 | 19
  Follow-Up Week 36 | 77.14 (18.25) | 72.37 (16.85)

3. Secondary Outcome: Asocial Belief Scale (ABS) Total Score
Description: Determine if CBSST + oxytocin compared to CBSST + placebo is associated with asocial beliefs. The total ABS score is calculated by adding the scores for items #1-#15. Each scale is provided a True/False response, with True responses equaling 1 point and False responses equaling 0 points. In calculating the ABS total score, four of the 15 items of the ABS were reverse scored. A lower total score indicates more severe asocial beliefs.
Time Frame: Treatment weeks 0, 12, and 24, plus follow-up week 36
Population: Only participants who were enrolled in the study and had completed a ABS assessment were analyzed at each study time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBSST + Oxytocin | CBSST + Placebo
Number analyzed (Participants) | 31 | 31
units on a scale
  Treatment Week 0 | 6.8 (3.6) | 5.5 (2.5)
  Treatment Week 12: number analyzed (Participants) | 27 | 24
  Treatment Week 12 | 6.8 (3.9) | 5.8 (3.1)
  Treatment Week 24: number analyzed (Participants) | 22 | 20
  Treatment Week 24 | 6.4 (2.8) | 5.2 (3.1)
  Follow-Up Week 36: number analyzed (Participants) | 21 | 19
  Follow-Up Week 36 | 6.6 (3.6) | 4.9 (3.2)

4. Secondary Outcome: Schedule for Assessment of Negative Symptoms (SANS) Total Score
Description: SANS total score range = 0-85. Higher scores indicate more severe negative symptoms.
Time Frame: Every 4 weeks during the treatment phase, plus follow-up week 36
Population: Only participants who were enrolled in the study and had completed a SANS assessment were analyzed at each study time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBSST + Oxytocin | CBSST + Placebo
Number analyzed (Participants) | 31 | 31
units on a scale
  Treatment Week 0 | 28.5 (12.5) | 35.9 (12.5)
  Treatment Week 4: number analyzed (Participants) | 29 | 25
  Treatment Week 4 | 25.3 (11.1) | 32.2 (10.6)
  Treatment Week 8: number analyzed (Participants) | 25 | 24
  Treatment Week 8 | 26.5 (10.9) | 30.8 (10.3)
  Treatment Week 12: number analyzed (Participants) | 26 | 24
  Treatment Week 12 | 26.0 (9.4) | 29.0 (11.8)
  Treatment Week 16: number analyzed (Participants) | 23 | 21
  Treatment Week 16 | 27 (8.5) | 30.7 (14.0)
  Treatment Week 20: number analyzed (Participants) | 20 | 21
  Treatment Week 20 | 25.5 (9.2) | 31.9 (14.2)
  Treatment Week 24: number analyzed (Participants) | 22 | 20
  Treatment Week 24 | 27.5 (9.5) | 31.2 (11.2)
  Follow-Up Week 36: number analyzed (Participants) | 22 | 20
  Follow-Up Week 36 | 27.1 (10) | 30.7 (11.3)

5. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) Total Score
Description: The total BPRS score is calculated by adding the scores for scales #1-#18. Each scale ranges from "1=Not Present" to "7=Very Severe". Total scores range from a minimum score of 18 to a maximum score of 126. A higher total score indicates a more severe psychiatric symptom rating.
Time Frame: Every 4 weeks during the treatment phase, plus follow-up week 36
Population: Only participants who were enrolled in the study and had completed a BPRS assessment were analyzed at each study time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBSST + Oxytocin | CBSST + Placebo
Number analyzed (Participants) | 31 | 31
units on a scale
  Treatment Week 0 | 38.2 (8.2) | 40.0 (10.4)
  Treatment Week 4: number analyzed (Participants) | 29 | 25
  Treatment Week 4 | 34.5 (6.7) | 39.1 (8.9)
  Treatment Week 8: number analyzed (Participants) | 25 | 24
  Treatment Week 8 | 33.5 (8.8) | 38.6 (9.2)
  Treatment Week 12: number analyzed (Participants) | 27 | 24
  Treatment Week 12 | 31.7 (6.0) | 37.9 (9.2)
  Treatment Week 16: number analyzed (Participants) | 23 | 21
  Treatment Week 16 | 30.5 (4.8) | 36.7 (10.5)
  Treatment Week 20: number analyzed (Participants) | 20 | 21
  Treatment Week 20 | 31.3 (7.0) | 37.2 (10.6)
  Treatment Week 24: number analyzed (Participants) | 22 | 20
  Treatment Week 24 | 33.7 (7.0) | 37.8 (9.8)
  Follow-Up Week 36: number analyzed (Participants) | 22 | 20
  Follow-Up Week 36 | 33.7 (5.9) | 39.0 (8.9)

6. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) Psychosis Score
Description: The psychosis score is calculated by adding the scores for scales #4 Conceptual Disorganization, #11 Suspiciousness, #12 Hallucinatory Behavior, and #15 Unusual Thought Content. Each scale ranges from "1=Not Present" to "7=Very Severe". The minimum psychosis score is 4 and the maximum psychosis score is 28. A higher score indicates a more severe psychosis rating.
Time Frame: Every 4 weeks during the treatment phase, plus follow-up week 36
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBSST + Oxytocin | CBSST + Placebo
Number analyzed (Participants) | 31 | 31
units on a scale
  Treatment Week 0 | 10.4 (4.9) | 11.7 (6.0)
  Treatment Week 4: number analyzed (Participants) | 29 | 25
  Treatment Week 4 | 9.7 (4.3) | 12.2 (5.7)
  Treatment Week 8: number analyzed (Participants) | 25 | 24
  Treatment Week 8 | 8.8 (3.7) | 12.9 (5.5)
  Treatment Week 12: number analyzed (Participants) | 27 | 24
  Treatment Week 12 | 7.7 (3.4) | 12.1 (5.0)
  Treatment Week 16: number analyzed (Participants) | 23 | 21
  Treatment Week 16 | 7.5 (3.0) | 11.0 (5.8)
  Treatment Week 20: number analyzed (Participants) | 20 | 21
  Treatment Week 20 | 8.3 (3.8) | 10.5 (5.7)
  Treatment Week 24: number analyzed (Participants) | 22 | 20
  Treatment Week 24 | 9.3 (3.9) | 11.2 (5.4)
  Follow-Up Week 36: number analyzed (Participants) | 22 | 20
  Follow-Up Week 36 | 8.8 (4.0) | 11.1 (5.2)

ADVERSE EVENTS:
Time Frame: Weekly for 24 weeks
Description: Reportable adverse events (AEs) are defined as any harm experienced by a study participant, which in the opinion of the investigator is unexpected and probably related to the research procedures. None of our AEs met these criteria.
  Participants are systematically monitored for any increases the Side Effects Checklist (SEC). An SEC AE includes any symptom/side effect rated with a score of 4 (severe) or for which there was a 2 point change in severity from baseline.
Arm/Group | CBSST + Oxytocin | CBSST + Placebo
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/31
Other Adverse Events (participants affected / at risk) | 3/31 | 5/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBSST + Oxytocin (N=31) | CBSST + Placebo (N=31)
Hospitalization (General disorders) | 1 (1) | 0 (0) — Hospitalization due to unrelated sinusitis
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — Hospitalization due to clinical worsening unrelated to study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBSST + Oxytocin (N=31) | CBSST + Placebo (N=31)
Dry mouth (General disorders) | 0 (0) | 2 (2)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Nasal irritation (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No